CLINICAL TRIAL: NCT01905449
Title: Biofeedback and Speech Disorders
Brief Title: Ultrasound Biofeedback for Speech Sound Disorders
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1303011662
Record Dates: First submitted 2013-07-16; First posted 2013-07-23 (Estimated); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Speech Sound Disorders
MeSH Terms: conditions — Speech Sound Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ultrasound plus prosodic cues (Experimental): One sound in error is treated with ultrasound visual feedback while also cueing prosodic variation (7 one-hour sessions). Another sound in error is treated with the ultrasound visual feedback with no prosodic variation (7 one-hour sessions). Prosodic variations are cues to coordinate production of the target sound with intonation patterns such as questions (rising intonations), commands (loud/emphatic), or statements (neutral)
  Interventions: Behavioral: Ultrasound visual feedback
- Ultrasound vs Traditional treatment (Experimental): One sound in errors is treated with ultrasound visual feedback for approximately half of each session and traditional treatment for half of the session (7 one-hour sessions). Another sound in error is treated with no ultrasound visual feedback, using traditional treatment for the entire session (7 one-hour sessions). These traditional cues include verbal instructions on how to move the tongue to achieve a particular speech sound.
  Interventions: Behavioral: Ultrasound visual feedback

INTERVENTIONS:
Behavioral: Ultrasound visual feedback — Real-time visual displays of the tongue are used to cue participants to modify the tongue position/shape as they articulate speech sounds

SUMMARY:
Children with speech sound disorders will receive speech therapy using real-time images of the tongue from ultrasound. These images will be used to cue the child to change the tongue position when producing speech sounds.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be native English-speaking children with no known hearing or vision deficits. Participants must be within the specified age range and have been identified as having speech production difficulties by a local speech-language therapist.

Exclusion Criteria:

* Participants will be excluded if there is a history of oral structural impairment (e.g., cleft palate), hearing or vision impairment, history of neurological impairment or injury, developmental disabilities such as Down Syndrome or Autism, or intellectual disability.

During initial testing, participants must score below a standard score of 75 on the Goldman-Fristoe Test of Articulation-2 and also score below 20% accurate on a probe list of words assessing accuracy of the /r/ sound

Ages: 8 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Actual)
Dates: Start 2013-05; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Percent correct for target speech sound | Change in accuracy after 7 one-hour treatment sessions (3.5 weeks), and after 14 one-hour treatment sessions (7 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Preston, PhD, Principal Investigator — Haskins Laboratories
Locations (1):
- Haskins Laboratories, New Haven, Connecticut, United States

REFERENCES:
- See also: Related Info — http://www.haskins.yale.edu/inner_content/studies.html